CLINICAL TRIAL: NCT04368494
Title: Exercise as an Anti-inflammatory Treatment in Axial Spondyloarthritis Patients (axSpA): a Proof of Concept Study (ExTASI).
Brief Title: Exercise Therapy in Patients With Axial Spondyloarthritis
Acronym: ExTASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Nicolette Bishop, Professor, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS project ID: 268333
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Axial Spondyloarthritis; Inflammatory Disease; Arthritis
Keywords: Exercise
MeSH Terms: conditions — Axial Spondyloarthritis; Arthritis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Random allocation into either a control group or an exercise group (12-weeks of home based exercise).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Continue with normal activity.
- Exercise (Experimental): 12-weeks of home based exercise involving 30 minutes of brisk walking on 5 days per week.
  Interventions: Behavioral: 12-week home based exercise

INTERVENTIONS:
Behavioral: 12-week home based exercise — Patients allocated to the exercise arm will be prescribed a home-based walking exercise programme consisting of 30 minutes of walking on 5 days per week at an RPE in the range of 12-14 (somewhat hard). Each patient's heart rate range will be established during the baseline exercise test by recording the heart rate response at the required RPE target range. This will be provided to each patient to use in conjunction with the activity monitor they will be given to wear on their non-dominant wrist. The monitor reports heart rate and records daily steps, distance and activity duration.
  Arms: Exercise

SUMMARY:
Regular exercise, such as brisk walking, has been shown to lower levels of indicators of inflammation in the blood in people with long term conditions. This includes people with heart disease, kidney disease and diabetes. Axial Spondyloarthritis (axSpA) is an inflammatory condition with prescribed medication focusing on reducing inflammation. However, the effect of exercise on indicators of inflammation in axSpA is unknown.

The research study intends to investigate whether a 12-week period of regular exercise can have favourable effects on inflammatory markers in the blood.

DETAILED DESCRIPTION:
Over 200,000 people in the UK have axial spondyloarthritis (axSpA). In 80% of cases the condition begins between 20-30 years of age. Exercise is encouraged as an essential treatment of axSpA, with the potential to promote well-being, flexibility, posture and pain management. Axial spondyloarthritis is an inflammatory arthritis and raised levels of indicators can be detected in the blood (e.g C-reactive protein). These markers are released as a consequence of the condition, but some, such as TNF-alpha, also promote further disease development.

In other patient groups with inflammatory diseases it has been demonstrated that regular exercise (brisk walking) can lower the levels of pro-inflammatory blood markers and increase levels of anti-inflammatory markers, independent of weight loss. Despite axSpA being an inflammatory condition with prescribed medication focused on reducing inflammation, there are no studies which have assessed the potential of exercise as an anti-inflammatory treatment in axSpA.

This research study will investigate the effect of 12 weeks of a home-based walking exercise intervention on measures of systemic inflammation and body composition. Measures of well-being and disease activity will also be investigated using established and validated methods. There will be an exercise and control group, both containing 10 participants. In the control group, patients will carry on with their normal activity. This proof-of-concept study will determine the potential of exercise as an additional anti-inflammatory treatment for patients with axSpA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Axial Spondyloarthritis by a consultant rheumatologist.
* Without other significant cardiovascular comorbidities.
* Receiving stable dose NSAID treatment.
* Able to commit to the time demands of the study.

Exclusion Criteria:

* Unable to undertake exercise due to physical or psychological barriers.
* Presence of hip or peripheral joint disease.
* Contraindication to exercise training (American College of Sports Medicine guidelines).
* Excessively active (score of high on International Physical Activity Questionnaire).
* Unable to communicate sufficiently in English.
* Female participants who are pregnant, lactating, or planning pregnancy during the course of the study.
* Inability to give informed consent or comply with the testing and training protocol for any reason.
* Presence of chronic anaemia.
* Co-morbidity that the research team determine to be a contraindication to involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in interleukin-6 blood concentrations before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Fasting blood concentration.
Changes in tumor necrosis factor-alpha blood concentrations before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Fasting blood concentration.
Changes in interleukin-10 blood concentrations before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Fasting blood concentration.
Changes in c-reactive protein blood concentrations before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Fasting blood concentration.

SECONDARY OUTCOMES:
Changes in creatine kinase blood concentrations before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Fasting blood concentration.
Changes in inflammatory immune cell phenotypes before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Expression of receptors associated with inflammatory activity and stimulated cell inflammatory cytokine release. This will be analysed via flow cytometry.
Changes in ankylosing spondylitis disease activity before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Using the validated Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The BASDAI consists of a 0-10 score (0 being no problem and 10 being the worst problem) which is used to answer 6 questions on fatigue, spinal pain, joint pain, tenderness, morning stiffness duration, and morning stiffness severity. To give each symptom equal weighting, the mean (average) of the two scores relating to stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score. The higher the score, the higher the activity of disease.
Changes in the symptom burden of ankylosing spondylitis before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Using the validated Bath Ankylosing Spondylitis Functional Index (BASFI). The index assesses the functional limitation in patients with anykylosing spondylitis by asking the patient about symptom burden. The index consists of 10 questions evaluating how hard the patient finds situations i.e 'how difficult is it to put on your socks?' A score of 0 represents easy, and a score of 10 represents impossible. The mean (average) of the 10 questions is used to assign a symptom burden score of 0-10. The higher the score, the higher the symptom burden caused by ankylosing spondylitis.
Changes in spinal pain before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Using the validated visual analogue scale for spinal pain. The scale consists of a straight line with the end points defining extreme limits 'no spinal pain' and 'spinal pain as bad as it could be'. The line is 10cm in length (0cm point representing no pain, 10cm point representing pain as bad as it could be). A score of 0-10 is given depending on where the patient marks the line (5cm representing a score of 5). The higher the score, the worse the spinal pain.
Changes in overall health status before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Using the validated Assessment of SpondyloArthritis Health Index (ASAS-HI). The health index assesses health in patients with spondyloarthritis. The questionnaire asks 17 questions to assess health, with a dichotomous response option: 'I agree' and 'I do not agree'. A score of 1 is given for each 'I agree' response, and a score of 0 is given for each 'I do not agree' response. The lower the total score, the better the overall health status.
Changes in work productivity before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Using the validated work productivity and activity impairment questionnaire (WPAI:GH). The questionnaire asks about the effect of health problems on the ability to work and perform regular activities. The questionnaire outcome is expressed as an impairment percentage, with higher numbers indicating greater impairment and less productivity.
Sedentary activity minutes per day | 7 days (+/- 3 days) in the 2 week period prior to baseline assessment.
  All participants will wear an Actigraph activity monitor on their non-dominant wrist to record physical activity for approximately 7 days (+/- 3 days) in the two weeks before the baseline assessment visit to characterise physical activity levels.
  The Freedson (1998) activity monitor counts per minute cut points will be used to quantify minutes per day spent sedentary.
Light physical activity minutes per day | 7 days (+/- 3 days) in the 2 week period prior to baseline assessment.
  All participants will wear an Actigraph activity monitor on their non-dominant wrist to record physical activity for approximately 7 days (+/- 3 days) in the two weeks before the baseline assessment visit to characterise physical activity levels.
  The Freedson (1998) activity monitor counts per minute cut points will be used to quantify minutes per day spent in light activity.
Moderate to vigorous physical activity minutes per day | 7 days (+/- 3 days) in the 2 week period prior to baseline assessment.
  All participants will wear an Actigraph activity monitor on their non-dominant wrist to record physical activity for approximately 7 days (+/- 3 days) in the two weeks before the baseline assessment visit to characterise physical activity levels.
  The Freedson (1998) activity monitor counts per minute cut points will be used to quantify minutes per day spent in moderate to vigorous physical activity.
Changes in subjective physical activity before (week 0 - baseline), during (week 12), and after (week 20) the 12-week home based exercise intervention. | 0, 12 and 20 weeks.
  Measured from the international physical activity questionnaire (IPAQ). The IPAQ asks 27 questions on physical activity (PA).
  Those who score 'high' engage in: 1) vigorous activity on at least 3 days achieving a total PA of at least 1500 metabolic equivalent of task (MET) minutes a week - OR - 2) 7 or more days of any combination of walking, moderate intensity or vigorous intensity activities achieving a minimum total PA of at least 3000 MET minutes per week.
  Those who score 'moderate' engage in: 1) 3 or more days of vigorous intensity activity and/or walking of at least 30 minutes per day - OR - 2) 5 or more days of moderate intensity activity and/or walking of at least 30 minutes per day - OR - 3) 5 or more days of any combination of walking, moderate intensity, or vigorous intensity activities achieving a minimum total PA of at least 600 MET minutes per week.
  Those who score 'low' do not fit the criteria of either the moderate or high levels of PA.
Changes in exercise tolerance before (week 0 - baseline), during (week 12), and after (week 20) the 12-week home based exercise intervention. | 0, 12 and 20 weeks.
  The participant will walk for 30 minutes on a motorised treadmill at a 1% gradient and at a speed that will elicit a perceived exertion of somewhat hard. The validated rating of perceiving exertion (RPE) scale will be used to quantify RPE. For the 30 minute duration, a combination of heart rate and rating of perceived exertion will be used to quantify exercise tolerance. A rating of perceived exertion of 6 represents no exertion, and a score of 20 represents maximal exertion. The score will be used to assess changes in exercise tolerance during (week 12) and after (week 20) the 12-week home based exercise intervention.
Changes in physical function before (week 0 - baseline), during (week 12), and after (week 20) the 12-week home based exercise intervention. | 0, 12 and 20 weeks.
  Sit to stand-5 test.
Changes in secondary physical function before (week 0 - baseline), during (week 12), and after (week 20) the 12-week home based exercise intervention. | 0, 12 and 20 weeks.
  Sit to stand-60 test.
Changes in height before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Centimetres
Changes in weight before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Kilograms
Changes in waist circumference before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Centimetres
Changes in hip circumference before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Centimetres
Changes in systolic blood pressure before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  mmHg.
Changes in diastolic blood pressure before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  mmHg.
Changes in body fat percentage before (week 0 - baseline), during (weeks 4, 8, and 12), and after (week 20) the 12-week home based exercise intervention. | 0, 4, 8, 12, 20 weeks.
  Via tanita body composition scales (bio electrical impedance analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Arumugam Moorthy, Dr, Principal Investigator — University Hospitals, Leicester
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester NHS trust, Leicester
  - Loughborough University, National Centre for Sport and Exercise Medicine, Loughborough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts MJ, Hamrouni M, Linsley V, Moorthy A, Bishop NC. Exercise as an anti-inflammatory Therapy in Axial Spondyloarthritis Therapeutic Intervention (EXTASI) study: a randomized controlled trial. Rheumatol Adv Pract. 2024 May 11;8(2):rkae062. doi: 10.1093/rap/rkae062. eCollection 2024. PMID 38854418